CLINICAL TRIAL: NCT05966870
Title: Reducing Added Sugar Intake on Sweetness Perception in Adolescents by Substituting Unsweetened Sparkling Water for Sugar Sweetened Beverages
Brief Title: Unsweetened Sparkling Water and Changes in Sweetness Perception in Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because this study was initiated during the COVID pandemic, several outcome measures (including those requiring in-person assessments) were abandoned.
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Nana Gletsu Miller, Associate Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1908757318; P30DK097512 (NIH)
Record Dates: First submitted 2023-07-10; First posted 2023-08-01 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Obesity, Adolescent; PreDiabetes
MeSH Terms: conditions — Pediatric Obesity; Prediabetic State

STUDY DESIGN:
Intervention Model Description: Prospective, before and after, cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Replacement of SSB with Unsweetened Sparkling Beverage (Experimental): To encourage participants to substitute sparkling water flavored water for SSB intake, we will provide enough supplies of the drinks to adolescents (and their families) each month. We will also provide iPhones with the TADA app to the adolescent participants. Study staff will remind participants to consume the sparkling water through iMessages sent through the TADA app.
  Interventions: Other: Unsweetened flavored sparkling water

INTERVENTIONS:
Other: Unsweetened flavored sparkling water — Unsweetened sparkling waters are carbonated water with flavoring, completely unsweetened, which are commercially available in soda-like flavors like cola

SUMMARY:
The study design is a prospective observational study in adolescents who are at risk for developing Type 2 Diabetes (T2D), to evaluate the effectiveness of sparkling water to reduce dietary intake of added sugars and thereby improve glycemia. Study data on consumption and the flavor profile of sparkling water will serve as a measure of acceptability. The study intervention will be to provide carbonated flavored sparkling water for 12 weeks to adolescents (and their families) who have a usual intake of 2 or more servings of sugar sweetened beverages (SSB) per day and are at a high risk for developing type 2 diabetes. Study measures will be obtained before and after the exposure to carbonated flavored sparkling water and each participant will serve as his/her own control. To encourage the participants to substitute the carbonated flavored sparkling water, study personnel will send them weekly iMessages through the Technology Assisted Dietary Assessment (TADA) app. In addition, investigators will monitor the participants' diet, using the TADA app, every two weeks, for 4 days. Study measurements will be obtained at baseline, before the intervention, during and at the end of the 12 week intervention.

Objective: Determine the effect of reducing added sugars intake by substituting carbonated sparkling water on T2D risk in adolescents.

Hypothesis: Adolescents who decrease consumption of SSB by substituting sparkling water will experience decreased blood glucose concentrations and increased insulin sensitivity during an oral glucose tolerance test and decreased glucose excursions during continued glucose monitoring, compared to those who do not decrease consumption of SSB.

DETAILED DESCRIPTION:
Importance of studying added sugars in adolescents. Research that leads to nutritional strategies to prevent T2D in adolescents is an urgent pursuit. One particular contributing factor to the growth of T2D and prediabetes in adolescents is the increased consumption of added sugars. Adolescents in the U.S. have high intakes of added sugars which could have poor health implications. Added sugars are found in sugar sweetened beverages and desserts and snacks, top sources of energy for adolescents, and calories from added sugars contribute to 16% of the total energy intake. Levels are well above recommendations from leading scientific organizations, which suggest limiting added sugars to less than 10% of energy. However, it is not clear whether sugar reduction to less than 10% of energy is palatable for an adolescent population that prefers sweetened foods and beverages. Moreover, uncertainty about the evidence linking added sugar consumption to risk of disease has made policies that seek to reduce dietary intake of added sugar controversial. The controversy impairs large-scale implementation of recommendations to reduce intake of added sugars by individuals, clinicians, policy makers and industry stakeholders.

Evidence linking added sugars and risk of type 2 diabetes and cardiovascular disease lacks information on adolescents. Many epidemiological studies in adults, but not all show the concept that after controlling for energy intake, high consumption of sugar-sweetened foods is a risk factor for T2D. Epidemiological studies also associate high consumption of added sugars, particularly from sugar sweetened beverages (SSB), with increased adiposity (including central adiposity) and dyslipidemia. These studies formed the basis of recommendations to limit added sugar consumption from the American Heart Organization. The data in youth is limited. Two small randomized studies compared the effects of glucose versus fructose beverages on insulin sensitivity in adolescents and findings were mixed. One longitudinal cohort study showed that higher consumption of added sugars, from SSB, was associated with hyperglycemia and impaired insulin sensitivity in youth aged 8 - 12 years. One study showed that high amounts of added sugars may induce insulin resistance and beta-cell dysfunction and such effects can occur independent of adiposity. The literature lacks evidence linking high consumption of added sugars to risk of developing youth-onset T2D.

Substituting Flavored Sparkling Water for Sugar Sweetened Beverages. Instead of sugar, food manufacturers typically sweeten foods beverages using low-calorie or artificial sweeteners. "Diet" versions of SSB have been available for several decades and are widely used by adults and children. However the safety of low calorie sweeteners is controversial and many in the scientific and lay communities do not promote their use as a substitute for SSB. We propose that an alternative to SSB may be found in sparkling waters (carbonated water with flavoring, completely unsweetened), which are commercially available in soda-like flavors like cola or Dr. Pepper™. The rationale for the current project is the urgent need for an effective strategy to combat adolescent T2D which investigators will address by demonstrating the benefit of an intervention to reduce added sugars. The objective of the study is to demonstrate whether substituting sparkling water for SSB has benefits for in vivo physiological measures of glycemia while maintaining flavor acceptability to adolescents who are at risk for diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adolescents (age 10-21 years)
* Overweight and Obese (body mass index ≥ 85 percentile for age and sex)
* High consumers of SSB, defined as >2 or more servings per day
* Family history of diabetes in a first or second degree relative OR prediabetes (i.e., evidence of either impaired glucose tolerance (HbA1c 5.7 - 6.4%, or plasma glucose between 140-199 mg/dL at 2 hours on oral glucose tolerance testing) or impaired fasting plasma glucose (≥ 100 mg/dL))

Exclusion Criteria:• Pregnancy

* Use of medications that affect glucose metabolism (such as glucocorticoid-containing medications or atypical antipsychotics). We will not exclude female participants who currently use, are planning to use, or planning to stop taking oral contraceptives.
* Syndromic obesity (such as Prader Willi, hypothalamic obesity, or Laurence-Moon-Biedl)

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — participant eligibility is based on self-representation of gender identity
Enrollment: 22 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nana Gletsu Miller, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Public Health, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andes LJ, Cheng YJ, Rolka DB, Gregg EW, Imperatore G. Prevalence of Prediabetes Among Adolescents and Young Adults in the United States, 2005-2016. JAMA Pediatr. 2020 Feb 1;174(2):e194498. doi: 10.1001/jamapediatrics.2019.4498. Epub 2020 Feb 3. PMID 31790544
- [Background] Banfield EC, Liu Y, Davis JS, Chang S, Frazier-Wood AC. Poor Adherence to US Dietary Guidelines for Children and Adolescents in the National Health and Nutrition Examination Survey Population. J Acad Nutr Diet. 2016 Jan;116(1):21-27. doi: 10.1016/j.jand.2015.08.010. Epub 2015 Sep 26. PMID 26391469
- [Background] Reedy J, Krebs-Smith SM. Dietary sources of energy, solid fats, and added sugars among children and adolescents in the United States. J Am Diet Assoc. 2010 Oct;110(10):1477-84. doi: 10.1016/j.jada.2010.07.010. PMID 20869486
- [Background] Bailey RL, Fulgoni VL, Cowan AE, Gaine PC. Sources of Added Sugars in Young Children, Adolescents, and Adults with Low and High Intakes of Added Sugars. Nutrients. 2018 Jan 17;10(1):102. doi: 10.3390/nu10010102. PMID 29342109
- [Background] Boushey CJ, Kerr DA, Wright J, Lutes KD, Ebert DS, Delp EJ. Use of technology in children's dietary assessment. Eur J Clin Nutr. 2009 Feb;63 Suppl 1(Suppl 1):S50-7. doi: 10.1038/ejcn.2008.65. PMID 19190645
- [Background] Running, C.A. Desensitization but not sensitization from commercial chemesthetic beverages. Food Quality and Preference 2018 Vol. 69 Pages 21-27; DOI: 10.1016/j.foodqual.2018.05.001
- [Background] Wang J, Light K, Henderson M, O'Loughlin J, Mathieu ME, Paradis G, Gray-Donald K. Consumption of added sugars from liquid but not solid sources predicts impaired glucose homeostasis and insulin resistance among youth at risk of obesity. J Nutr. 2014 Jan;144(1):81-6. doi: 10.3945/jn.113.182519. Epub 2013 Nov 6. PMID 24198307
- [Background] Matsuda M, DeFronzo RA. Insulin sensitivity indices obtained from oral glucose tolerance testing: comparison with the euglycemic insulin clamp. Diabetes Care. 1999 Sep;22(9):1462-70. doi: 10.2337/diacare.22.9.1462. PMID 10480510

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Started | 22
Completed | 11
Not Completed | 11

BASELINE CHARACTERISTICS:
Population: Demographic summary of study participants that completed the 12-week intervention
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: years] | 19.9 [10 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Dietary Consumption of SSB and Sparkling Water
Description: Dietary consumption of SSB and Sparkling water were assessed using Technology Assisted Dietary Assessment (TADA) system, a mobile food record
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: Because we were unable to complete in-person training due to the COVID pandemic, there was poor adoption of the TADA system during the COVID-19 pandemic, and valid/sufficient data collection was not completed for any of the participants.
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 0

2. Primary Outcome: Change in 2 Hour Glucose Concentrations
Description: Oral glucose tolerance testing will be performed in the morning after participants have undergone an overnight fast for 8 hours at baseline and Week 12. Blood samples will be obtained at -15, 0, 15, 30, 60, 90,120 minutes, relative to ingestion of a glucose drink at a dose of 1.75 g/kg body weight (maximum 75 g glucose).
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: Because of the COVID-19 pandemic, data were not collected for this outcome measure (as in-person assessments were abandoned).
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 0

3. Primary Outcome: Change in Fasting Glucose
Description: Fasting glucose will be measured after overnight fast for 8 hours, just prior to the initiation of the baseline oral glucose tolerance testing at Baseline and Week 12.
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 2
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 0

4. Primary Outcome: Change in Hemoglobin A1c (HbA1c) Concentration
Description: HbA1c will be measured just prior to the initiation of the oral glucose tolerance testing at baseline and Week 12.
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 2
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 0

5. Primary Outcome: Change in Whole-body Insulin Sensitivity Index (WBISI)
Description: For measures of insulin action, which takes into account serum glucose and insulin concentrations, serum fractions from the oral glucose tolerance tests will be frozen at -80 degrees C until analysis. The inverse of fasting insulin (1/fasting insulin) will be used as a surrogate estimate of whole-body insulin sensitivity.
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 2
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 0

6. Primary Outcome: Change in Insulinogenic Index (IGI)
Description: For measures of insulin action, which takes into account serum glucose and insulin concentrations, serum fractions from the oral glucose tolerance tests will be frozen at -80 degrees C until analysis. Early phase insulin secretion during the OGTT will be expressed as the insulinogenic index (IGI) or the ratio of the incremental response of insulin to glucose at 30 minutes of the OGTT (IGI30).
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 2
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 0

7. Primary Outcome: Change in Oral Disposition Index (oDI)
Description: For measures of insulin action, which takes into account serum glucose and insulin concentrations, serum fractions from the oral glucose tolerance tests will be frozen at -80 degrees C until analysis. The oDI will be calculated as IGI30 × 1/fasting insulin.
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 2
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 0

8. Primary Outcome: Change in Glycemic Control
Description: We will collect free-living, glucose measures for 6 consecutive days using the Continuous Glucose Monitoring (CGM; FreeStyle Libre Pro System; Abbott; Abbott Park, IL). The CGM will be administered to participants 6 days before the start of Week 0 and Week 12, and the monitor will be removed at the clinic visit. For the placement of the CGM, the back of the participant's upper arm will be cleaned with an alcohol wipe and dried. The sensor will be firmly adhered to the arm with the needle application inserted. The FreeStyle sensor measures glucose every 15 sec and records an average glucose value every 15 min for up to 14 days.
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 2
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 0

9. Secondary Outcome: Change in Flavor Perception of Beverage Sweetness - Tested With a Beverage With Sugar Concentration 0% (Weight Per Volume)
Description: Participants consumed a test beverage with sugar concentration 0% (weight per volume), and rated the beverage using a "Just About Right" (JAR) visual analog scale for sweetness perception. The JAR scale anchors at: -100, "Not sweet enough"; -50, "Slightly not sweet enough"; 0, "Just about right"; +50, "Slightly too sweet"; and +100 "Too sweet." In this scale, the greater the deviation from zero the more suboptimal the perception.
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: The analysis population included all participants who completed both the pre- and post-intervention assessments, measured per JAR scale.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 11
score on a scale
  JAR pre intervention | -90 [-95 to -20]
  JAR post intervention | -75 [-90 to -25]

10. Secondary Outcome: Change in Flavor Perception of Beverage Sweetness - Tested With a Beverage With Sugar Concentration 1.8% (Weight Per Volume)
Description: Participants consumed a test beverage with sugar concentration 1.8% (weight per volume), and rated the beverage using a "Just About Right" (JAR) visual analog scale for sweetness perception. The JAR scale anchors at: -100, "Not sweet enough"; -50, "Slightly not sweet enough"; 0, "Just about right"; +50, "Slightly too sweet"; and +100 "Too sweet." In this scale, the greater the deviation from zero the more suboptimal the perception.
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 9
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 11
score on a scale
  JAR pre intervention | -50 [-95 to -30]
  JAR post intervention | -20 [-95 to 0]

11. Secondary Outcome: Change in Flavor Perception of Beverage Sweetness - Tested With a Beverage With Sugar Concentration 2.8% (Weight Per Volume)
Description: Participants consumed a test beverage with sugar concentration 2.8% (weight per volume), and rated the beverage using a "Just About Right" (JAR) visual analog scale for sweetness perception. The JAR scale anchors at: -100, "Not sweet enough"; -50, "Slightly not sweet enough"; 0, "Just about right"; +50, "Slightly too sweet"; and +100 "Too sweet." In this scale, the greater the deviation from zero the more suboptimal the perception.
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 9
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 11
score on a scale
  JAR pre intervention | -5 [-45 to 0]
  JAR post intervention | 0 [-50 to 30]

12. Secondary Outcome: Change in Flavor Perception of Beverage Sweetness - Tested With a Beverage With Sugar Concentration 4.4% (Weight Per Volume)
Description: Participants consumed a test beverage with sugar concentration 4.4% (weight per volume), and rated the beverage using a "Just About Right" (JAR) visual analog scale for sweetness perception. The JAR scale anchors at: -100, "Not sweet enough"; -50, "Slightly not sweet enough"; 0, "Just about right"; +50, "Slightly too sweet"; and +100 "Too sweet." In this scale, the greater the deviation from zero the more suboptimal the perception.
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 9
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 11
score on a scale
  JAR pre intervention | -10 [-50 to 50]
  JAR post intervention | 5 [-45 to 60]

13. Secondary Outcome: Change in Flavor Perception of Beverage Sweetness - Tested With a Beverage With Sugar Concentration 6.8% (Weight Per Volume)
Description: Participants consumed a test beverage with sugar concentration 6.8% (weight per volume), and rated the beverage using a "Just About Right" (JAR) visual analog scale for sweetness perception. The JAR scale anchors at: -100, "Not sweet enough"; -50, "Slightly not sweet enough"; 0, "Just about right"; +50, "Slightly too sweet"; and +100 "Too sweet." In this scale, the greater the deviation from zero the more suboptimal the perception.
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 9
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 11
score on a scale
  JAR pre intervention | 30 [-5 to 100]
  JAR post intervention | 60 [5 to 100]

14. Secondary Outcome: Change in Flavor Perception of Beverage Sweetness - Tested With a Beverage With Sugar Concentration 10.7% (Weight Per Volume)
Description: Participants consumed a test beverage with sugar concentration 10.7% (weight per volume), and rated the beverage using a "Just About Right" (JAR) visual analog scale for sweetness perception. The JAR scale anchors at: -100, "Not sweet enough"; -50, "Slightly not sweet enough"; 0, "Just about right"; +50, "Slightly too sweet"; and +100 "Too sweet." In this scale, the greater the deviation from zero the more suboptimal the perception.
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 9
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 11
score on a scale
  JAR pre intervention | 60 [-5 to 100]
  JAR post intervention | 80 [65 to 95]

15. Secondary Outcome: Change in Hedonic Visual Scale for Liking - Tested With a Beverage With Sugar Concentration 0% (Weight Per Volume)
Description: Participants consumed a test beverage with sugar concentration 0% (weight per volume) and rated the beverage for liking using a hedonic visual analog scale. This scale anchors at: -100, "Worst ever"; -50, "Dislike"; 0, "Neutral"; +50, "Like"; +100, "Best ever".
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: The analysis population included all participants who completed both the pre- and post-intervention assessments using the hedonic visual analog scale for liking
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 11
score on a scale
  Liking rating pre intervention | -45 [-95 to 10]
  Liking rating post intervention | 7 [-55 to 55]

16. Secondary Outcome: Change in Hedonic Visual Scale for Liking - Tested With a Beverage With Sugar Concentration 1.8% (Weight Per Volume)
Description: Participants consumed a test beverage with sugar concentration 1.8% (weight per volume) and rated the beverage for liking using a hedonic visual analog scale. This scale anchors at: -100, "Worst ever"; -50, "Dislike"; 0, "Neutral"; +50, "Like"; +100, "Best ever".
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 15
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 11
score on a scale
  Liking rating pre intervention | 0 [-67 to 100]
  Liking rating post intervention | 45 [-4 to 100]

17. Secondary Outcome: Change in Hedonic Visual Scale for Liking - Tested With a Beverage With Sugar Concentration 2.8% (Weight Per Volume)
Description: Participants consumed a test beverage with sugar concentration 2.8% (weight per volume) and rated the beverage for liking using a hedonic visual analog scale. This scale anchors at: -100, "Worst ever"; -50, "Dislike"; 0, "Neutral"; +50, "Like"; +100, "Best ever".
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 15
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 11
score on a scale
  Liking rating pre intervention | 25 [-45 to 80]
  Liking rating post intervention | 50 [-55 to 70]

18. Secondary Outcome: Change in Hedonic Visual Scale for Liking - Tested With a Beverage With Sugar Concentration 4.4% (Weight Per Volume)
Description: Participants consumed a test beverage with sugar concentration 4.4% (weight per volume) and rated the beverage for liking using a hedonic visual analog scale. This scale anchors at: -100, "Worst ever"; -50, "Dislike"; 0, "Neutral"; +50, "Like"; +100, "Best ever".
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 15
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 11
score on a scale
  Liking rating pre intervention | 20 [-60 to 80]
  Liking rating post intervention | 30 [-30 to 80]

19. Secondary Outcome: Change in Hedonic Visual Scale for Liking - Tested With a Beverage With Sugar Concentration 6.8% (Weight Per Volume)
Description: Participants consumed a test beverage with sugar concentration 6.8% (weight per volume) and rated the beverage for liking using a hedonic visual analog scale. This scale anchors at: -100, "Worst ever"; -50, "Dislike"; 0, "Neutral"; +50, "Like"; +100, "Best ever".
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 15
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 11
score on a scale
  Liking rating pre intervention | 50 [-75 to 100]
  Liking rating post intervention | 25 [-30 to 100]

20. Secondary Outcome: Change in Hedonic Visual Scale for Liking - Tested With a Beverage With Sugar Concentration 10.7% (Weight Per Volume)
Description: Participants consumed a test beverage with sugar concentration 10.7% (weight per volume) and rated the beverage for liking using a hedonic visual analog scale. This scale anchors at: -100, "Worst ever"; -50, "Dislike"; 0, "Neutral"; +50, "Like"; +100, "Best ever".
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 15
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 11
score on a scale
  Liking rating pre intervention | 30 [-65 to 97]
  Liking rating post intervention | 35 [-70 to 70]

21. Secondary Outcome: Change in Blood Triglycerides
Description: Plasma triglyceride concentration will be measured.
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 2
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 0

22. Secondary Outcome: Change in Blood Pressure
Description: Blood pressure will be measured after 5 minutes of rest, on the right arm in the supine position.
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 2
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 0

23. Secondary Outcome: Change in Waist Circumference
Description: The distance around the waist will be measured.
Time Frame: Between 0 and 12 weeks (pre-testing was at week 0, post-testing at week 12)
Population: as for outcome 2
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: During the 12 week study
Description: Any change in the health condition of the participants
Arm/Group | Replacement of SSB With Unsweetened Sparkling Beverage
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

LIMITATIONS AND CAVEATS:
Because of the Covid-19 pandemic, data were not collected for the following outcomes:

* Change in Dietary consumption of SSB and Sparkling water assessed with the TADA system
* 2 hour Glucose Concentrations Measured Using 2 hour Oral Glucose Tolerance Testing
* Fasting glucose and Hemoglobin A1C
* Insulin Sensitivity measures (WBISI, IGI, and oDI)
* Glycemic Control Measured Using Continuous Glucose Monitoring
* CVD Outcomes (Blood Triglycerides, Blood Pressure and Waist Circumference)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT05966870/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT05966870/SAP_001.pdf